CLINICAL TRIAL: NCT00365469
Title: A Follow-up Study to 5 Years of a Randomized, Double-blinded, Placebo-controlled Study on the Influence of Probiotics on Atopy, Immunological Responses and Gut Microflora
Brief Title: Influence of Probiotics on Atopy, Immunological Responses and Gut Microflora - Follow-up to 5 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Paediatrics, Dr Marion Aw, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SQNU01 (Phase II)
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2014-01

CONDITIONS: Eczema; Asthma; Allergic Rhinitis
Keywords: Probiotics; Eczema; Asthma; Allergic Rhinitis; Prevention; Immunological responses
MeSH Terms: conditions — Eczema; Asthma; Rhinitis, Allergic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic (Experimental): Commercially available cow's milk based infant formula with Bifidobacterium longum [BL999} and Lactobacillus rhamnosus [LPR]
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Commercially available cow's milk based infant formula without probiotic supplementation
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Bifidobacterium longum [BL999] and Lactobacillus rhamnosus [LPR]
  Arms: Probiotic
Other: Placebo — Commercially available cow's milk based infant formula without probiotic supplementation
  Arms: Placebo

SUMMARY:
The investigators had conducted a double-blind, randomized placebo-controlled clinical trial studying the effects of 6 months probiotics supplementation from birth on allergic disease and sensitization up to 2 years of age. This follow-up study will extend a further 3 years to 5 years of age for assessing the longer term beneficial effects of this form of probiotics intervention on the incidence of allergic disease and sensitization at 5 years of age.

DETAILED DESCRIPTION:
Probiotics are helpful bacteria of healthy gut and have shown potential in reducing allergy. A double-blind, randomized placebo-controlled clinical trial studying the effects of 6 months probiotics supplementation from birth on allergic disease and sensitization up to 2 years of age had been conducted. This study aims to assess the longer term beneficial effects of this form of intervention on the incidence of allergic disease and sensitization at 5 years of age by extending the follow-up period.

All children (from original cohort of 253) who completed the initial 2-year visit has been invited to participate. They will be evaluated with monthly phone calls and yearly clinic visits. Allergic sensitization will be assessed with skin prick tests to a panel of allergens.

This project will provide insights into the role of early supplementation of probiotics on the development of the immune system and its effect on allergy. The additional follow-up period is critical for the evaluation of respiratory allergies in the form of clinical asthma, allergic rhinitis and sensitization to inhalant allergens, which tend to develop after 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Parents agree to the subject's participation in the study and informed consent has been obtained.
* The subject has been a participant in the Phase I double-blind, randomized placebo-controlled study and had taken either normal infant formula or formula supplemented with probiotics postnatally for 6 months.
* The parents are willing to comply with study procedures and are able to keep to scheduled clinic visits.

Exclusion Criteria:

* The parent is unable /unwilling to comply with procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2006-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Asthma | 5 years of age

SECONDARY OUTCOMES:
Atopic eczema | 5 years of age
Allergic Rhinitis | 5 years of age
Allergen sensitization | 5 years of age
Food Allergy | 5 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marion Aw, Consultant, Principal Investigator — National University Hospital, Singapore; Dr Lynette Shek, Consultant, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore